CLINICAL TRIAL: NCT00871091
Title: Pilot Study Investigating Tooth Movements With Conventional and CAD/CAM Supported Fixed Appliances
Brief Title: Study Investigating Tooth Movements With Conventional and Computer-Aided Design/Computer-Aided Manufacturing (CAD/CAM) Supported Fixed Appliances
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Charite University, Berlin, Germany (Other)
Collaborators: German Research Foundation (Other)
Responsible Party: Paul-G. Jost-Brinkmann, Prof. Dr., Charité - Universitätsmedizin Berlin
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: JO 207/4-1-4
Record Dates: First submitted 2009-03-27; First posted 2009-03-30 (Estimated); Last update posted 2009-03-30 (Estimated); Status verified 2009-03

CONDITIONS: Tooth Movement; Orthodontics
Keywords: CAD/CAM; orthodontics; fixed appliance; tooth movement
MeSH Terms: interventions — Orthodontics

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- 1 (Experimental): CAD/CAM group, customized archwires
  Interventions: Procedure: orthodontic treatment with customized archwires
- 2 (Active Comparator): prefabricated archwires (superelastic)
  Interventions: Procedure: orthodontic treatment with prefabricated archwires
- 3 (Active Comparator): prefabricated archwires with manual adjustments
  Interventions: Procedure: orthodontic tx w/ conventional archwires+manual adjustments

INTERVENTIONS:
Procedure: orthodontic treatment with customized archwires — customized arch wires depending on the amount of needed tooth movement
  Other Names: SureSmile; CAD/CAM
  Arms: 1
Procedure: orthodontic treatment with prefabricated archwires — prefabricated archwires depending of the needed movement of the teeth
  Other Names: archwires, prefabricated; conventional orthodontic treatment
  Arms: 2
Procedure: orthodontic tx w/ conventional archwires+manual adjustments — conventional archwires modified by manual adjustment, depending of needed correction
  Other Names: manual adjustment; conventionel archwires
  Arms: 3

SUMMARY:
In orthodontics, conventional fixed appliances, usually consisting of prefabricated components, require step-by-step adjustment in order to move teeth in the planned direction.

May treatment be improved with customized archwires?

Study hypotheses:

* By using CAD/CAM in planning and fabrication of customized archwires, unnecessary tooth movements can be avoided and teeth can be moved on their direct path to the intended position.
* The application of CAD/CAM improves reproducibility, efficiency, and quality of orthodontic treatment.

ELIGIBILITY:
Inclusion Criteria:

* treatment of front teeth with fixed orthodontic appliances is indicated
* complete secondary dentition
* age: 18-35
* in healthy general condition
* patient is informed about study and agrees to participate

Exclusion Criteria:

* treatment of premolars and molars is necessary
* syndromes affecting bones and teeth
* cleft lip and palate
* inflammation or reduction (more than 50%) of periodontium
* intake of drugs affecting tooth movement and bone formation
* disturbance of bone formation
* disturbance of thyroidal function
* pregnancy
* participation in additional study affecting oral hygiene
* former therapy with ionized radiation or cytostatic drugs
* caries (active phase)
* alcohol dependency

Ages: 18 Years to 35 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 32 (Estimated)
Dates: Start 2007-01; Primary Completion 2009-05 (Estimated); Study Completion 2009-06 (Estimated)

PRIMARY OUTCOMES:
Sum of differences between resulted and shortest path of tooth movements in each patient | measurements every 14 days until end of treatment

SECONDARY OUTCOMES:
Difference between resulted and shortest path of movements for each tooth | measurements every 14 days until end of treatment

CONTACTS AND LOCATIONS:
Overall Officials: Paul-Georg Jost-Brinkmann, Prof, Study Chair — Charite - Universitätsmedizin
Locations (1):
- Department of Orthodontics, Dentofacial Orthopedics and Pedodontics, Charité - Universitätsmedizin Berlin, Berlin, Germany